CLINICAL TRIAL: NCT01158846
Title: Bivalirudin Plus Prasugrel vs Abciximab Plus Clopidogrel. Optimizing Ischemic Protection and Bleeding Risk in Patients With ST Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Bivalirudin/Prasugrel Versus Abciximab/Clopidogrel in Patients Presenting With STEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: Centro Cardiologico Monzino (Other); Azienda Ospedaliera Niguarda Cà Granda (Other); Istituto Clinico Humanitas (Other)
Responsible Party: Dr. Luca Testa, Istituto Clinico S.Ambrogio
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Biva/Pra versus Abcix/clop; B/P vs A/C for STEMI (Registry Identifier: Milan STEMI registry); Biva/Pra versus Abcix/clop (Registry Identifier: Biva/Pra versus Abcix/clop); Biva/Pra versus Abcix/clop (Registry Identifier: Milan STEMI registry)
Record Dates: First submitted 2010-06-25; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-06

CONDITIONS: ST-Elevation Myocardial Infarction; Primary Percutaneous Coronary Intervention
Keywords: STEMI; Primary PCI; anticoagulants; antiplatelets
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride; bivalirudin; Clopidogrel; Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prasugrel/bivalirudin (Active Comparator): 60 mg loading dose of prasugrel will be followed by maintenance dose of 10mg (or 5mg according to body weight and age). During primary PCI, Bivalirudin will be used as anticoagulant (bolus plus infusion), on a weight-adjusted dose.
  Interventions: Drug: prasugrel/bivalirudin
- clopidogrel/abciximab (Active Comparator): 600mg loading dose of clopidogrel will be followed by 75mg maintenance dose. During primary PCI abciximab (bolus plus infusion) will be used as anticoagulant.
  Interventions: Drug: clopidogrel/abciximab

INTERVENTIONS:
Drug: prasugrel/bivalirudin — 60mg loading dose followed by 10mg or 5 mg (according to body weight or age)maintenance dose of prasugrel. Bivalirudin during the primary PCI (bolus plus infusion)
  Other Names: Efient; Angiox
  Arms: prasugrel/bivalirudin
Drug: clopidogrel/abciximab — 600mg loading dose of clopidogrel followed by 75mg maintenance dose. Abciximab will be used during primary PCI, bolus plus infusion.
  Other Names: Plavix; ReoPro
  Arms: clopidogrel/abciximab

SUMMARY:
In the setting of ST elevation myocardial infarction newer therapies has been recently studied and, following encouraging results, introduced into the clinical practice. Prasugrel showed to be a valid alternative to overcome limitation of clopidogrel therefore providing a better ischemic protection. On the other hand, bivalirudin is at least as beneficial as heparin/abciximab as anticoagulant agent but associated with fewer hemorrhagic events. The primary hypothesis of the study is that the combination of prasugrel plus bivalirudin can be associated with a better risk/benefit profile.

DETAILED DESCRIPTION:
Background:

In the setting of STEMI, adjunctive pharmacological therapy plays a key role in the acute management. Along with the clear benefit of mechanical reperfusion strategies, several drugs showed to be beneficial. On top of clopidogrel, heparins and IIB/IIIa glycoprotein, other drugs have been recently introduced showing encouraging results. These "new" drugs, namely prasugrel and bivalirudin, have only been compared separately.

Primary hypothesis: the combination of prasugrel/bivalirudin is superior to the combination of clopidogrel and heparin/abciximab in terms of net adverse clinical events, i.e. ischemic events plus hemorrhagic events

Setting:

- patients presenting with ST-elevation myocardial infarction undergoing primary PCI

Mechanical reperfusion:

-primary percutaneous coronary intervention

Pharmacological Interventions:

- Two arms: Clopidogrel plus heparin/abciximab vs Prasugrel plus Bivalirudin

Follow up:

- 1 year

Measurements:

* efficacy end points in terms of reduction of ischemic events
* safety end points in terms of reduction of bleeding events

ELIGIBILITY:
Inclusion Criteria:

* ST elevation myocardial infarction
* No contraindication to primary PCI

Exclusion Criteria:

* Known intolerance/allergy to one of the study drugs or their components
* Clinical indication to treatment with oral anticoagulant, including use of warfarin or dabigatran or other oral anticoagulant agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 1 year
  Combined outcome of overall death, non fatal MI, major stroke

SECONDARY OUTCOMES:
major bleedings | 1 year
  according to TIMI major bleedings definition
minor bleedings | 1 year
  according to TIMI minor bleedings definition
stent thrombosis | 1 year
  according to ARC definition of probable/definite stent thrombosis
overall death | 1 year
non fatal myocardial infarction | 1 year
  defined according to current guidelines
ischemic stroke | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Luca Testa, MD,PhD, Principal Investigator — Istituto Clinico S. Ambrogio; Fracensco Bedogni, MD, Study Director — Istituto Clinico S. Ambrogio
Locations (1):
- Istituto Clinico S. Ambrogio, Milan, Italy

REFERENCES:
- [Background] Montalescot G, Wiviott SD, Braunwald E, Murphy SA, Gibson CM, McCabe CH, Antman EM; TRITON-TIMI 38 investigators. Prasugrel compared with clopidogrel in patients undergoing percutaneous coronary intervention for ST-elevation myocardial infarction (TRITON-TIMI 38): double-blind, randomised controlled trial. Lancet. 2009 Feb 28;373(9665):723-31. doi: 10.1016/S0140-6736(09)60441-4. PMID 19249633
- [Background] Mehran R, Lansky AJ, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Gersh BJ, Pocock SJ, Wong SC, Nikolsky E, Gambone L, Vandertie L, Parise H, Dangas GD, Stone GW; HORIZONS-AMI Trial Investigators. Bivalirudin in patients undergoing primary angioplasty for acute myocardial infarction (HORIZONS-AMI): 1-year results of a randomised controlled trial. Lancet. 2009 Oct 3;374(9696):1149-59. doi: 10.1016/S0140-6736(09)61484-7. Epub 2009 Aug 28. PMID 19717185